CLINICAL TRIAL: NCT02435004
Title: Clinical Study Protocol Dorsal Root Ganglion Stimulation for the Management of Painful Intractable Small Fibre Neuropathy
Brief Title: Dorsal Root Ganglion Stimulation for the Management of Painful Intractable Small Fibre Neuropathy:
Acronym: NSI-TD-002
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Regionale di Lugano (Other)
Responsible Party: Principal Investigator, Eva Koetsier MD PhD LLM, MD PhD LLM, Ospedale Regionale di Lugano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSI-TD-002
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Neuropathy Small Fibre
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Modulation Axium™ (Other): Spinal Modulation Axium™: an external trial neurostimulator (TNS) is used for the trial period, followed by an implanted neurostimulator (INS) if the TNS is successful. The TNS and INS are a pacemaker-sized devices that send out mild electrical pulses. The stimulator contains a battery and electrical components. Both TNS and INS are constant voltage devices. The TNS is used first and is worn on the outside of the clothing. The INS is implanted under the skin and support:
  Interventions: Device: Spinal Modulation Axium™

INTERVENTIONS:
Device: Spinal Modulation Axium™ — The participants will undergo implantation of electrodes for stimulation of fuor dorsal ganglia (Spinal Modulation, Inc., Menlo Park, CA, USA). Each participant will have one to four electrodes positioned according to the individual distribution of pain in the extremities. After implantation the electrode will be connected to an external neurostimulator: Spinal Modulation Axium™ for 3-30 days to evaluate their effectiveness (test stimulation).
  If during the trial treatment the pain will decrease significantly (> 50%) a neurostimulator will be 'implanted for the continuation of the permanent neurostimulation. The neurostimulator is implanted in the abdomen in a subcutaneous pocket.

SUMMARY:
A prospective, single-arm, mono-centre pilot study to obtain preliminary information on the ability of Dorsal Root Ganglion Stimulation (DRGS) in alleviating the painful symptoms in patients with small fiber neuropathy (SFN).

DETAILED DESCRIPTION:
This study is a prospective, single-arm, mono-centre pilot study enrolling a maximum of 31 patients with SFN. All enrolled patients will receive a trial neurostimulation (TNS) lasting from 3 to 30 days and only patients with a positive result in terms of pain intensity reduction will be eligible for the implanted neurostimulation (INS) phase. The target number of patients eligible for INS is 10 and this population will be assessed for impact of DRGS on the neuropathic pain caused by SFN. The expected duration of patients participation will be 14 months. The rationale for this open label approach is that this is a novel technique for which pilot data with regard to applicability and efficacy have yet to be established. Data gathered in the study will provide preliminary data required to assess the feasibility of this intervention, to be used for possible future studies with a more rigorous methodological approach (i.e. controlled trial, randomized controlled trial).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at inclusion
* Chronic, intractable painful SFN in the peripheral limbs during at least 12 months and a biopsy positive for SFN, with a chronic pain intensity of ≥ 6 on a Numeric Rating Scale (ranging from 0 to 10), for which previous drug therapy was unsuccessful
* Stable medication dosage in the 30 days prior to inclusion
* Stable pattern of neurological symptoms

Exclusion Criteria:

* Known or suspected non-compliance
* Drug or alcohol abuse
* Pain predominantly in upper limbs
* Neuropathy or chronic pain in limbs of other origin than SFN
* Peripheral vascular disease
* Severe foraminal stenosis at the expected target level
* Coagulation disorders
* Known immune-deficiency
* Other significant concomitant diseases and any concomitant malignancies
* Presence of other indwelling devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-04; Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity assessed by Numeric Rating Scale. | Pain intensity assessment during 2 weeks after inmplatation, at Time point 6 and 12 months after implantation.
  Four assessments/day for 5 consecutive days around the intended measurement timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- EOC Lugano, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Koetsier E, Vacchi E, Maino P, Dukanac J, Melli G, van Kuijk SMJ. Dorsal Root Ganglion Stimulation in Chronic Painful Polyneuropathy: A Potential Modulator for Small Nerve Fiber Regeneration. Neuromodulation. 2023 Dec;26(8):1772-1780. doi: 10.1016/j.neurom.2022.08.455. Epub 2022 Oct 1. PMID 36192280